CLINICAL TRIAL: NCT05040126
Title: Evaluate the Effectiveness, Safety and Tolerability of Various Doses of Linezolid in Combination With Bedaquiline and Pretomanid in Adults With Pre-Extensively Drug-Resistant (Pre-XDR), Or Treatment Intolerant/Non-responsive Multidrug-Resistant (MDRTI/NR) Pulmonary Tuberculosis in India
Brief Title: Modified BPaL Regimen for Managing Pre-XDR TB and MDR (TI/NR) TB in India
Acronym: mBPaL
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tuberculosis Research Centre, India (Other Government)
Collaborators: International Union Against Tuberculosis and Lung Diseases (Other); Sarvodaya Charitable Trust Hospital, Ghatkopar, Mumbai (Unknown); Shatabdi Centenary Hospital, Govandi, Mumbai (Unknown); King George's Medical College and Hospital, Lucknow (Unknown); SN Medical College, Agra (Unknown); Govt Medical College & Hospital, Bhavnagar (Unknown); Govt. Medical College & Hospital, Surat (Unknown); National Institute for Tuberculosis and Respiratory Diseases, New Delhi (Unknown); Rajan Babu Institute of Pulmonary Medicine and Tuberculosis, Delhi (Unknown); Govt.Rajaji Medical college and hospital, Madurai (Unknown)
Responsible Party: Principal Investigator, Dr C Padmapriyadarsini, Director, Tuberculosis Research Centre, India
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021 004
Record Dates: First submitted 2021-08-18; First posted 2021-09-10 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Pre-Extensively Drug-Resistant Pulmonary TB; Treatment Intolerant Multidrug-Resistant Pulmonary TB; Non-responsive Multidrug-Resistant Pulmonary TB
MeSH Terms: interventions — Linezolid; bedaquiline; pretomanid

STUDY DESIGN:
Intervention Model Description: Pragmatic Clinical Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1 - 26 weeks of BDQ +Pa + LZD (600mg) (Active Comparator): 26 wks. of BDQ +Pa + LZD (600mg) Bedaquiline (available as 100 mg tablets) Bedaquiline will be administered as four 100 mg tablets (400 mg) by mouth once a day for 2 weeks, followed by two 100 mg tablets (200 mg) by mouth three times a week for 24 weeks.
  Linezolid: (available as 600 mg tablets) - Linezolid will be administered as one 600 mg tablet once daily in Arm1.
  Pretomanid: (Available as 200 mg tablets): Pretomanid is administered as one tablet once a day for 26 weeks along with Bedaquiline and Linezolid.
  Interventions: Drug: Linezolid; Drug: Bedaquiline; Drug: Pretomanid
- Arm 2 - 9 weeks. of BDQ +Pa + LZD (600mg) followed by 17 wks. of BDQ +Pa+ LZD (300mg) (Experimental): 9 wks. of BDQ +Pa + LZD (600mg) followed by 17 wks. of BDQ +Pa+ LZD (300mg) Bedaquiline (available as 100 mg tablets) Bedaquiline will be administered as four 100 mg tablets (400 mg) by mouth once a day for 2 weeks, followed by two 100 mg tablets (200 mg) by mouth three times a week for 24 weeks.
  Linezolid: (available as 600 mg tablets) - Linezolid will be administered as one 600 mg tablet once daily in IP of Arm 2 and ½ tablet of 600 mg once daily in CP of Arm 2 .
  Pretomanid: (Available as 200 mg tablets): Pretomanid is administered as one tablet once a day for 26 weeks along with Bedaquiline and Linezolid.
  Interventions: Drug: Linezolid; Drug: Bedaquiline; Drug: Pretomanid
- Arm 3 -13 weeks. of BDQ +Pa + LZD (600mg) followed by 13 wks. of BDQ +Pa+ LZD (300mg) (Experimental): 13 wks. of BDQ +Pa + LZD (600mg) followed by 13 wks. of BDQ +Pa+ LZD (300mg) Bedaquiline (available as 100 mg tablets) Bedaquiline will be administered as four 100 mg tablets (400 mg) by mouth once a day for 2 weeks, followed by two 100 mg tablets (200 mg) by mouth three times a week for 24 weeks.
  Linezolid: (available as 600 mg tablets) - Linezolid will be administered as one 600 mg tablet once daily in IP of Arm 3 and ½ tablet of 600 mg once daily in CP of Arm 3.
  Pretomanid: (Available as 200 mg tablets): Pretomanid is administered as one tablet once a day for 26 weeks along with Bedaquiline and Linezolid.
  Interventions: Drug: Linezolid; Drug: Bedaquiline; Drug: Pretomanid

INTERVENTIONS:
Drug: Linezolid — Participants will have a screening period of up to 14 days and will be randomized to one of the study arms in the ratio of 1:1:1, using an interactive web response system.
  Each participant will receive 26 weeks of treatment. If the participant's 16th-week sample remains culture positive, treatment will be extended up to 39 weeks.
  Participants will be followed for 48 weeks after the end of treatment
Drug: Bedaquiline — Bedaquiline will be administered as four 100 mg tablets (400 mg) by mouth once a day for 2 weeks, followed by two 100 mg tablets (200 mg) by mouth three times a week for 24 weeks in all three arms
Drug: Pretomanid — Pretomanid is administered as one tablet once a day for 26 weeks in all three arms

SUMMARY:
Existing problem with DR TB management:

Injectable regimens for longer duration with toxicity Poor adherence, treatment failures, continued transmission

Need of the study:

Oral regimens of shorter duration Improved treatment adherence Implementation of community-based models of care Reduction in direct costs and indirect costs of patients Improved treatment outcomes

Need for shorter, tolerable and effective regimen

Hence modified BPaL regimen is designed to study the newer shorter oral in varying doses of Linezolid for pre XDR Tb patients and MDR TI/NR patients

DETAILED DESCRIPTION:
The regimen proposed is based on the NIX-TB and ZeNIX trial regimen with modification in the Linezolid doses. The rationale is -

1. While the EBA study showed that a modestly greater bactericidal effect over 14 days at the highest 1200 mg daily, this dose appears to be associated with a greater incidence of neuropathic and myelosuppressive effects than the 600 mg daily dose in the NIXTB trial.
2. Linezolid EBA study showed similar bactericidal activity over 14 days irrespective of the single daily dose or twice-daily doses. A single daily dose will enhance patient adherence and will reduce the total time of exposure to the drug concentration that is greater than the calculated concentration associated with mitochondrial toxicity (likely mechanism for the toxicities of peripheral neuropathy and myelosuppression).
3. While a full 6 months of linezolid therapy in the regimen may give greater culture conversion and avoid relapse, the mouse model found that linezolid dosing only for one or two months, when B and Pa were given continuously for a total of 3 months, maximized relapse-free cure.
4. More than 2 months of linezolid, when combined with B and Pa, does not increase relapse-free cure in the mouse model. Thus, the treatment arms in this study will give randomized comparative information about the optimal duration and dose of linezolid in the regimen relative to efficacy and toxicity.
5. The ZeNIX study with consistent dosing of bedaquilline and pretomanid reported 93% success rate with linezolid 1200 mg for 6 months and 91% with linezolid 600mg for 6 months. However 2 months of 600mg linezolid showed a success rate of 84%. Adverse reactions were reported in 38 % of those receiving 1200mg linezolid for 6 months, 24% of those receiving 600mg of linezolid for 6 months and 13% of those receiving 600mg linezolid for 2 months.
6. Interim analysis of BEAT study (personal communication/52nd UNION abstract) with 6 month regimen of bedaquilline, delaminid, clofazimine and linezolid (600mg daily for 6 months) reported 89.6% success rate at the end of 6 months of treatment. Adverse reactions such as peripheral neuropathy were reported in 39% and myelosuppression in 47% of the patients.

Learning from ZeNIX and BEAT study, a planned reduction of Linezolid along with BDQ and Pretomanid is planned as BDQ+Pa+LZD 600mg for 9 weeks followed by 300 mg for 17 weeks and BDQ+Pa+LZD 600mg for 13 weeks followed by 300mg for 13 weeks. This will help in deciding the effective dosing of Lzd to be combined with Bdq and Pa for drug resistant TB in the program.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged between 18 years - 65 years
2. Pulmonary Pre-XDR-TB, patients [with documented evidence of resistance to rifampicin with or without isoniazid resistance AND additional resistance to any fluoroquinolones by conventional DST (culture-based1) or rapid DST (Xpert MTB/RIF or Trunat MTB/RIF or LPA) from a certified laboratory] OR MDR-TBTI/NR patients [with documented treatment intolerance or non-response to MDR TB treatment regimen for 6-months or more when the participant was adherent to the treatment regimen]
3. Bodyweight of ≥30 kg (in light clothing and no shoes)
4. Provide written, informed consent before all study-related procedures
5. Provide consent to HIV testing2 (if an HIV test was performed within 1 month before the study start, it should not be repeated as long as documentation can be provided [ELISA and/or Western Blot]).
6. Aspartate aminotransferase (AST) or Alanine aminotransferase (ALT) < 2.5 x ULN; Total bilirubin lesser than ULN when accompanied by an increase in other liver function tests.
7. QTcF less than or equal to 450 at baseline
8. Female patients should not be pregnant or should be using a birth control method. They should be willing to continue practicing birth control methods (barrier or non-barrier contraceptive methods including oral contraceptives) throughout the treatment period, or history of post-menopausal for the past 12 months.

Exclusion Criteria:

Non-DST based criteria

1. Intolerance or risk of toxicity from medicine in the treatment regimens (e.g. drug-drug interactions)
2. Patient who has received more than 2 weeks of Bedaquiline or Linezolid before the first dose of BPaL regimen
3. Pregnancy or Lactating women
4. All forms of Extrapulmonary TB (Lymph node TB associated with Pulmonary DR-TB and pleural effusion associated with pulmonary TB can be considered for inclusion )
5. HIV infected patient having a CD4+ cell count of ≤ 50 cells/µL;
6. Currently having an uncontrolled cardiac arrhythmia that requires medication
7. Have any of the following QTcF interval characteristics at screening:

   1. QTcF ≥ 450 at baseline & normal electrolytes, ECG to be repeated after 6 hours and if both ECGs show QTc>450 then the patient should not be challenged with cardiotoxic drugs.
   2. History of additional risk factors for Torsade de Pointes, e.g. heart failure, hypokalaemia, family history of long QT syndrome;
8. Any condition in the Investigator's opinion (i.e., an unstable disease such as uncontrolled diabetes on insulin3 or cardiomyopathy), where participation would compromise the well-being of the patient or prevent, limit or confound protocol-specified assessments.
9. Very seriously ill patients (Karnofsky scores < 50 within last 30 days)
10. If results of the serum chemistry panel or, hematology are outside the normal reference range (as given below), the patient may still be considered if the physician judges that the abnormalities or deviations from normal to be not clinically significant or to be appropriate and reasonable.

    * Hypokalaemia, hypomagnesemia, and hypocalcemia should be corrected before a patient receiving any cardiotoxic drugs. (hypothyroidism is not exclusion criteria, to be considered with simultaneous thyroxine replacement therapy and close monitoring)
    * Haemoglobin level of < 9.0 g/dl or Platelet count <1,00,000 /mm3
    * Aspartate aminotransferase (AST) or Alanine aminotransferase (ALT) >2.5 x ULN; Total bilirubin greater ULN when accompanied by an increase in other liver function tests
11. Grade III or IV peripheral neuropathy

DST based criteria

a. if the result for DST (FQ, LZD)4 is not available and h/o more than 2 weeks consumption of drugs used in the study regimen

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-10-07 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Sustained Treatment success | 12 months after successful TB treatment
  Sustained Treatment success at 12 months after successful TB treatment, who is alive and free of TB. Successful TB treatment includes Cure and Treatment Completed.

SECONDARY OUTCOMES:
Proportion of serious adverse events | treatment and follow-up period - 18 months
  1. Proportion of serious adverse events occurring among patients in the study during the treatment and follow-up period
proportion of patients died | treatment and follow-up period - 18 months
  Died due to any cause during treatment
proportion of patients with Treatment Failure | treatment and follow-up period - 18 months
  Treatment terminated or need for permanent regimen change to a new regimen or treatment strategy because of lack of sputum culture conversion , • bacteriological reversion , clinical or radiological worsening
proportion of patients with Lost-to-follow up | treatment and follow-up period - 18 months
  After treatment initiation, treatment was interrupted continuously for 30-days

OTHER OUTCOMES:
HRQoL scores | baseline, end of treatment, and 48-weeks post-treatment - 18 months
  percentage change in score over the treatment period between the regimens

CONTACTS AND LOCATIONS:
Overall Officials: Padmapriyadarsini Chandrasekharan, Principal Investigator — Tuberculosis Research Centre, India
Locations (1):
- S N Medical College, Agra, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Padmapriyadarsini C, Devaleenal B, Ponnuraja C, Ramraj B, Singla R, Parmar M, Mattoo S, Mandal S. Randomised trial to evaluate the effectiveness and safety of varying doses of linezolid with bedaquiline and pretomanid in adults with pre-extensively drug-resistant or treatment intolerant/non-responsive multidrug-resistant pulmonary tuberculosis: study protocol. BMJ Open. 2022 Aug 29;12(8):e058606. doi: 10.1136/bmjopen-2021-058606. PMID 36038181